CLINICAL TRIAL: NCT05421169
Title: Invasive funCtional assEssment Using Diastolic HypEremia-Free RATio in Patient With Coronary Artery Disease: a Prospective Observation Study (ICE-HEAT)
Brief Title: Diastolic Hyperemia-Free Ratio in Patients With CAD
Acronym: ICE-HEAT
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Yongcheol Kim, Clinical Associate Professor, Yonsei University
Other Study IDs: 9-2022-0047
Record Dates: First submitted 2022-06-05; First posted 2022-06-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Coronary Stenosis; Coronary Artery Disease
Keywords: coronary artery disease; FFR; DFR
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: diastolic hyperemia-free ratio (DFR) — diastolic hyperemia-free ratio uses the mean Pd/Pa calculated over the period in diastole defined as that during which arterial pressure is negatively sloped and below the mean arterial pressure

SUMMARY:
The investigators aimed to identify the value of concordance between the diastolic hyperemia-free ratio (DFR) and fractional flow reserve (FFR) during pre-interventional and post-interventional period using a 0.014" COMET II Pressure Guidewire

DETAILED DESCRIPTION:
The physiologic assessment of coronary artery disease and ischemia-guided percutaneous coronary intervention (PCI) has become a standard practice for patients with coronary artery disease. Fractional flow reserve (FFR) represents hyperemic flow limitation caused by an epicardial coronary stenosis and its clinical usefulness has been proven by many clinical studies. However, the FFR is limited to clinical use despite the fact that it is recommended by the guideline due to the inconvenience of patients using medications used to induce maximum hyperemia, and the need for additional procedure time. Recently, a physiologic index which does not require hyperemia, instantaneous wave free ratio (iFR), was introduced and recent trials showed non-inferiority of iFR-guided strategy for 1-year clinical outcome, compared with FFR-guided strategy. Recently, not only iFR but also various intravascular pressure measurement techniques have been developed, one of which is diastolic hyperemia-free ratio (DFR). DFR uses the mean Pd/Pa calculated over the period in diastole defined as that during which arterial pressure is negatively sloped and below the mean arterial pressure. DFR showed equivalence as compared to gold standard FFR in the discrimination of non-culprit lesions requiring revascularization in patients with NSTEMI. In the case of DFR, there is no issue in terms of safety because it is conducted in the same way as iFR, but there are not many studies on the validation between DFR and FFR. Therefore, the present study aimed to identify the quality of concordance between DFR and FFR, determine the features associated with discrepancies in DFR and FFR.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ≥ 19 years of age, who are diagnosed with stable angina pectoris including silent ischemic heart disease and 50~90% stenosis of the coronary artery.
* Acute coronary syndrome patients with multivessel disease who have 50~90% stenosis of a non-culprit vessel on coronary angiography.

Exclusion Criteria:

* Patients with acute coronary syndrome and single vessel disease.
* Patients with hypersensitivity or contraindication to antiplatelet treatment.
* Female of childbearing potential, who possibly plan to become pregnant any time after enrollment into this study.
* Patients with a life expectancy shorter than 1 year.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients of stable angina pectoris including silent ischemic heart disease and 50~90% stenosis of coronary artery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Comparison of pre-interventional value between DFR <=0.89 and FFR <=0.80 | through study completion, an average of 1 year
  Efficacy and correlation of two invasive indexes of functional assessment by intracoronary pressure guidance in intermediate lesions with a cut-off point to defer the treatment of FFR< = 0.80 (with intravenous sigmart) and DFR < = 0.89.

SECONDARY OUTCOMES:
Comparison of the value between DFR <=0.89 and Pd/Pa <=0.92 | through study completion, an average of 1 year
  Efficacy and correlation of two invasive indexes of functional assessment by intracoronary pressure guidance in intermediate lesions with a cut-off point to defer the treatment of and DFR < = 0.89 and Pd/Pa <=0.92.
  Pd/Pa (resting distal to aortic coronary pressure) was evaluated as the ratio of mean aortic pressure (Pa) to mean distal coronary arterial pressure (Pd), After getting the Pd/Pa value, investigators performed DFR computation considering average Pd/Pa during the period between Pa less than mean Pa ending at systole and calculated using auto-mated algorithms (Boston scientific) acting during a minimum of three beats.
Comparison of post-interventional value between DFR >=0.89 and FFR >=0.80 when DFR/FFR-guided PCI is performed. | through study completion, an average of 1 year
  When the patients refered to PCI due to FFR <=0.80 or DFR <=0.89 for coronary stenotic lesion, investigators compared with post-interventional value between DFR and FFR after PCI.
Comparison of the delta value (Δ post-interventional - pre-interventional value) between DFR and FFR. | through study completion, an average of 1 year
  When PCI will be conduced, the comparison of the delta value between pre and post value of DFR and FFR will be measured.
Discordance factors between DFR >=0.89 and FFR >=0.80 | through study completion, an average of 1 year
  After assessment of DFR and FFR, the investigators collected the date of mismatch between DFR >=0.89 and FFR >=0.80 and analyzed the discordance factors between DFR >=0.89 and FFR >=0.80
Mortality within 30 days | through study completion, an average of 1 year
  umber of participants who died due to sudden cardiac arrest, sudden death due to acute MI and death due to heart failure or cardiogenic shock within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Principal Investigator — Yongin Severance Hopistal
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Roh JW, Lee OH, Kim Y, Heo SJ, Im E, Cho DK. Diastolic Hyperemia-Free Ratio in Patients With Coronary Artery Disease: A Prospective Observational Study. Korean Circ J. 2025 Jul;55(7):600-610. doi: 10.4070/kcj.2024.0351. Epub 2025 Feb 17. PMID 40206008